CLINICAL TRIAL: NCT05765266
Title: ACP Max™ PRP System for Knee Osteoarthritis: A Feasibility Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIRR-0032
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study where subjects and evaluators are blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ACP Max™ (Experimental): Single 4-6 ml intra-articular (IA) injection of the output of ACP Max™
  Interventions: Device: ACP Max™
- 40 mg of methylprednisolone acetate (Active Comparator): Single IA injection of 40 mg of methylprednisolone acetate (1 ml of solution) mixed with 5 ml of Normal Saline for a total of 6 ml.
  Interventions: Device: Depo-Medrol®

INTERVENTIONS:
Device: ACP Max™ — Single 4-6 ml intra-articular (IA) injection of the output of ACP Max™
  Arms: ACP Max™
Device: Depo-Medrol® — Single IA injection of 40 mg of methylprednisolone acetate (1 ml of solution) mixed with 5 ml of Normal Saline for a total of 6 ml.
  Other Names: methylprednisolone acetate)
  Arms: 40 mg of methylprednisolone acetate

SUMMARY:
This study is a prospective, multicenter (up to 4 sites), randomized, double-blind, two-arm study. Forty-five (45) patients will be randomized to receive a single 4-6 ml intra-articular (IA) injection of either the output of ACP Max™ (n=30) or 6 ml of Depo-Medrol® (methylprednisolone acetate) (n=15).

DETAILED DESCRIPTION:
All subjects will have a screening visit and a treatment visit followed by six follow-up visits: 10 days, 6 weeks, 3 months, 6 months, 9 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily decides to participate and signs the consent form.
2. Subject is ≥ 18 to 75 years of age.
3. Subject presents with symptomatic knee OA despite at least 6 months of one of the following conservative treatments; oral medications, analgesics, and/or anti-inflammatory medications.
4. Subject has documented radiographic evidence of OA in the tibiofemoral or patellofemoral compartment of the target knee (Kellgren-Lawrence Grades II-III), using radiographs performed within 12 weeks of screening.
5. Subject has a WOMAC pain score (WOMAC A) of at least 8 out of 20 and at least moderate degree of difficulty (a score of 2) for at least 2 questions on performing daily activities.
6. Subject consents to a washout period of NSAIDs and analgesics 7 days before each study visit (except low-dose aspirin for prevention of cardiovascular disease).
7. Subject has a Body Mass Index ≤ 35 kg/m2

Exclusion Criteria:

1. Subject has Grade I or IV in the target knee according to the Kellgren-Lawrence grading scale.
2. Subject has clinically 3+ effusion of the target knee (stroke test grading system).
3. Subject has significant (> 10°) valgus or varus deformities as evidenced by standard of care x-ray.
4. Subject has received an IA injection of corticosteroids in the target knee within 4 months prior to screening.
5. Subject did not achieve initial pain relief from prior corticosteroid injections.
6. Subject has received an IA injection of HA in the target knee within 6 months prior to screening.
7. Subject has received an IA injection of PRP in the target knee at any time prior to screening.
8. Subject has a history of coagulopathy.
9. Subject has joint pain reflected by a VAS score of > 35 mm out of 100 mm scale in the contralateral knee at the time of screening.
10. Subject had prior open surgery on the target knee within 12 months or knee arthroscopy within 6 months.
11. Subject has an inflammatory disease of either knee other than OA.
12. Subject which, in the investigator's opinion, has an underlying medical condition(s) that could interfere with the evaluation of the outcome.
13. Subject with a positive pregnancy test or breastfeeding.
14. Subject plans to participate in other clinical trials involving medical or surgical intervention in the next 12 months.
15. Subject with any condition (including cognitive impairment) that, in the investigator's opinion, might interfere with the evaluation of the study objectives.
16. Subject has rheumatoid arthritis or gout.
17. Subject has an infection at the affected joint.
18. Subject has a history of major trauma to the target knee within one year.
19. Subject with plans to undergo any elective orthopedic surgery in the next 12 months.
20. Subject requires pain management therapy not related to the target knee (with the exception of acetaminophen).
21. Subject has a known hypersensitivity to Depo-Medrol and its constituents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  A comparison of the frequency and severity of all adverse events between the investigational group and the control group at 6 months.
Adverse Events | 12 months
  Analysis of the frequency and severity of all adverse events for the investigational group at 12 months.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Likert Scale | Day 10, 6 weeks, 3, 6, 9 and 12 Months
  A 24-item questionnaire with 3 subscales measuring pain, stiffness, function and total scores.
Medication Usage | Day 10, 6 weeks, 3, 6, 9 and 12 months
  Medication Usage related to knee pain.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - AMR Knoxville, Knoxville, Tennessee
  - Spectrum Medical, Inc., Danville, Virginia

IPD SHARING:
Plan to Share IPD: No